CLINICAL TRIAL: NCT01901146
Title: A Randomized, Double-Blind, Phase 3 Study Evaluating the Efficacy and Safety of ABP 980 Compared With Trastuzumab in Subjects With HER2 Positive Early Breast Cancer
Brief Title: Efficacy and Safety Study of ABP 980 Compared With Trastuzumab in Women With HER2-positive Early Breast Cancer
Acronym: Lilac
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120283; 2012-004319-29 (EudraCT Number)
Record Dates: First submitted 2013-05-20; First posted 2013-07-17 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: Human Epidermal Growth Factor Receptor 2 (HER2); Positive Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Mastectomy, Segmental; Mastectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABP 980 (Experimental): Participants received ABP 980 at an initial dose of 8 mg/kg by intravenous (IV) infusion, then 6 mg/kg IV infusion every 3 weeks (Q3W) for 3 additional cycles plus 175 mg/m² paclitaxel Q3W for 4 cycles during the neoadjuvant phase.
  Surgery (lumpectomy or mastectomy with sentinel lymph node dissection or axillary lymph node dissection) was completed 3 to 7 weeks after the last dose of study drug in the neoadjuvant phase.
  After surgery (adjuvant phase) participants continued receiving 6 mg/kg ABP 980 IV Q3W for up to 1 year from the first day of study drug administration in the neoadjuvant phase.
  Interventions: Drug: ABP 980; Drug: Paclitaxel; Procedure: Lumpectomy or Mastectomy with Sentinel Node or Axillary Node Dissection
- Trastuzumab (Active Comparator): Participants received trastuzumab at an initial dose of 8 mg/kg IV infusion, then 6 mg/kg IV infusion Q3W for 3 additional cycles plus 175 mg/m² paclitaxel Q3W for 4 cycles during the neoadjuvant phase.
  Surgery (lumpectomy or mastectomy with sentinel lymph node dissection or axillary lymph node dissection) was completed 3 to 7 weeks after the last dose of study drug in the neoadjuvant phase.
  After surgery (adjuvant phase) participants were re-randomized to either continue receiving 6 mg/kg trastuzumab IV Q3W or transition to 6 mg/kg ABP 980 IV Q3W for up to 1 year from the first day of study drug administration in the neoadjuvant phase.
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Procedure: Lumpectomy or Mastectomy with Sentinel Node or Axillary Node Dissection

INTERVENTIONS:
Drug: ABP 980 — ABP 980 was administered at an initial dose of 8 mg/kg over a 90-minute intravenous (IV) infusion, then 6 mg/kg IV infusion Q3W for all subsequent cycles.
  Arms: ABP 980
Drug: Trastuzumab — Trastuzumab was administered at an initial dose of 8 mg/kg over a 90-minute IV infusion, then 6 mg/kg IV infusion Q3W for all subsequent cycles.
  Other Names: Herceptin®
  Arms: Trastuzumab
Drug: Paclitaxel — Paclitaxel, 175 mg/m² Q3W for 4 cycles (or 80 mg/m² QW for 12 cycles, if local standard of care).
Procedure: Lumpectomy or Mastectomy with Sentinel Node or Axillary Node Dissection

SUMMARY:
The purpose of this research study is to compare the effectiveness and safety of ABP 980 against trastuzumab in women with human epidermal growth factor receptor 2 (HER2)-positive early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥ 18 years of age
* Histologically confirmed invasive breast cancer
* Planning for surgical resection of breast tumor and sentinel node or axillary lymph node resection
* Planning neoadjuvant chemotherapy
* HER2 positive disease
* Measurable disease in the breast after diagnostic biopsy, defined as longest diameter ≥ 2.0 cm
* Known estrogen receptor (ER) and progesterone receptor (PR) hormone receptor status at study entry
* Normal bone marrow function
* Normal hepatic function
* Normal renal function
* Subjects must sign an Institutional Review Board/Ethics Committee (IRB/EC)-approved informed consent form before any study specific procedures

Inclusion Criteria for Randomization:

* Left ventricular ejection fraction (LVEF) of ≥55% by 2D echocardiogram
* Complete all 4 cycles of run-in chemotherapy

Exclusion Criteria:

* Bilateral breast cancer
* Presence of known metastases
* Received prior treatment, including chemotherapy, biologic therapy, radiation or surgery with the exception of diagnostic biopsy for primary breast cancer
* Other concomitant active malignancy or history of malignancy in the past 5 years except treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Pre-existing clinically significant (≥ grade 2) peripheral neuropathy
* Any history of documented or current congestive heart failure, current high-risk uncontrolled arrhythmias, current angina pectoris requiring a medicinal product, current clinically significant valvular disease, current evidence of transmural infarction on electrocardiogram (ECG), or current poorly controlled hypertension
* Severe dyspnea at rest requiring supplementary oxygen therapy
* History of positivity for hepatitis B surface antigen, hepatitis C virus, or human immunodeficiency virus (HIV)
* Recent infection requiring a course of systemic anti-infectives that were completed ≤ 14 days before enrollment (with the exception of uncomplicated urinary tract infection)
* Woman of childbearing potential who is pregnant or is breast feeding
* Woman of childbearing potential who is not consenting to use highly effective methods of birth control (eg, true abstinence [periodic abstinence (eg calendar ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception], sterilization, or other non-hormonal forms of contraception) during treatment and for at least 7 months after the last administration of the protocol specified treatment
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study
* Other investigational procedures while participating in this study are excluded
* Subject has known sensitivity to any of the products to be administered during the study, including mammalian cell derived drug products, trastuzumab, murine proteins, or to any of the excipients
* Subject previously has enrolled and/or has been randomized in this study
* Subject likely to not be available to complete all protocol required study visits or procedures
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the Investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Actual)
Dates: Start 2013-04-29 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (87):
- Belarus (3):
  - Research Site, Brest
  - Research Site, Grodno
  - Research Site, Minsk
- Brazil (6):
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Ijuí, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Jaú, São Paulo
  - Research Site, Santo André, São Paulo
  - Research Site, São Paulo, São Paulo
- Bulgaria (4):
  - Research Site, Sofia, Sofia
  - Research Site, Veliko Tarnovo, Veliko Tarnovo
  - Research Site, Pleven
  - Research Site, Varna
- Canada (2):
  - Research Site, Moncton, New Brunswick
  - Research Site, Montreal, Quebec
- Chile (2):
  - Research Site, Temuco, Cautín
  - Research Site, Santiago
- Germany (5):
  - Research Site, Fürstenwalde, Brandenburg
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Bonn, North Rhine-Westphalia
  - Research Site, Bottrop, North Rhine-Westphalia
  - Research Site, Berlin
- Greece (3):
  - Research Site, Athens, Attica
  - Research Site, Heraklion, Crete
  - Research Site, Thessaloniki, Nea Efkarpia
- Hungary (5):
  - Research Site, Debrecen, Hajdú-Bihar
  - Research Site, Szolnok, Jász-Nagykun-Szolnok
  - Research Site, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Research Site, Szekszárd, Tolna County
  - Research Site, Budapest
- Italy (7):
  - Research Site, San Fermo della Battaglia, COMO
  - Research Site, Bari
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, Piacenza
  - Research Site, Varese
- Mexico (4):
  - Research Site, Toluca, Estado de Mexico, Mexico
  - Research Site, Monterrey, Nuevo León
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Querétaro
- Poland (6):
  - Research Site, Poznan, Greater Poland Voivodeship
  - Research Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Research Site, Warszawa, Lublin Voivodeship
  - Research Site, Warsaw, Masovian Voivodeship
  - Research Site, Gdansk, Pomeranian Voivodeship
  - Research Site, Rybnik, Silesian Voivodeship
- Romania (5):
  - Research Site, Cluj-Napoca, Cluj
  - Research Site, Ploieşti, Prahova
  - Research Site, Timișoara, Timiș County
  - Research Site, Brasov
  - Research Site, Cluj-Napoca
- Russia (12):
  - Research Site, Obninsk, Kaluzhskaya
  - Research Site, Moscow Region, Moscow
  - Research Site, Arkhangelsk, Primorskiy (Maritime) Kray
  - Research Site, Saransk, Respublika Mordoviya
  - Research Site, Yaroslavl, Yaroslavlr
  - Research Site, Chelaybinsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Pyatigorsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Sochi
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
- South Africa (3):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Cape Town, Western Cape
- Spain (6):
  - Research Site, Sabadell, Barcelona
  - Research Site, A Coruña, LA Coruna
  - Research Site, Lleida, Lleida
  - Research Site, Alcorcón, Madrid
  - Research Site, Barcelona
  - Research Site, Madrid
- Ukraine (8):
  - Research Site, Kyiv, Kyiv City
  - Research Site, Lutsk, Volyn Oblast
  - Research Site, Uzhhorod, Zakarpattia Oblast
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Kharkiv
  - Research Site, Lviv
  - Research Site, Zaporizhzhya
- United Kingdom (2):
  - Research Site, Nottingham, England
  - Research Site, Peterborough, England

REFERENCES:
- [Derived] Kolberg HC, Colleoni M, Demetriou GS, Santi P, Tesch H, Fujiwara Y, Tomasevic Z, Hanes V. Cardiac Safety of the Trastuzumab Biosimilar ABP 980 in Women with HER2-Positive Early Breast Cancer in the Randomized, Double-Blind, Active-Controlled LILAC Study. Drug Saf. 2020 Mar;43(3):233-242. doi: 10.1007/s40264-019-00886-3. PMID 31927716
- [Derived] von Minckwitz G, Colleoni M, Kolberg HC, Morales S, Santi P, Tomasevic Z, Zhang N, Hanes V. Efficacy and safety of ABP 980 compared with reference trastuzumab in women with HER2-positive early breast cancer (LILAC study): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2018 Jul;19(7):987-998. doi: 10.1016/S1470-2045(18)30241-9. Epub 2018 Jun 4. PMID 29880292
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 123 sites in 20 countries from April 2013 to January 2017. The study consisted of a neoadjuvant treatment phase for 4 cycles, surgery, and adjuvant treatment for up to one year from the first day of study drug administration in the neoadjuvant phase.
Pre-assignment Details: Enrolled patients received run-in chemotherapy consisting of epirubicin and cyclophosphamide every 3 weeks for 4 cycles. After the run-in, participants with adequate cardiac function were randomized. Randomization was stratified by tumor stage, nodal status, hormone receptor status, planned paclitaxel dosing schedule, and geographic region.
Groups:
- ABP 980: Participants received ABP 980 at an initial dose of 8 mg/kg over a 90-minute intravenous (IV) infusion, then 6 mg/kg IV infusion every 3 weeks (Q3W) for 3 additional cycles plus 175 mg/m² paclitaxel Q3W for 4 cycles.
- Trastuzumab: Participants received trastuzumab at an initial dose of 8 mg/kg over a 90-minute IV infusion, then 6 mg/kg IV infusion Q3W for 3 additional cycles plus 175 mg/m² paclitaxel Q3W for 4 cycles.
- ABP 980/ABP 980: After surgery, participants initially randomized to ABP 980 continued to receive ABP 980 at a dose of 6 mg/kg IV infusion Q3W for up to 1 year from the first day of study drug administration in the neoadjuvant phase.
- Trastuzumab/Trastuzumab: After surgery, participants originally randomized to trastuzumab were re-randomized and continued to receive trastuzumab at a dose of 6 mg/kg IV infusion Q3W for up to 1 year from the first day of study drug administration in the neoadjuvant phase.
- Trastuzumab/ABP 980: After surgery, participants originally randomized to trastuzumab were re-randomized and switched to receive ABP 980 at a dose of 6 mg/kg IV infusion Q3W for up to 1 year from the first day of study drug administration in the neoadjuvant phase.
Period: Neoadjuvant Phase
Arm/Group | ABP 980 | Trastuzumab | ABP 980/ABP 980 | Trastuzumab/Trastuzumab | Trastuzumab/ABP 980
Started | 364 | 361 | 0 | 0 | 0
Completed | 358 (Indicates participants who completed surgery) | 347 (Indicates participants who completed surgery) | 0 | 0 | 0
Not Completed | 6 | 14 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 0 | 0 | 0
Not completed — Disease Progression or Recurrence | 2 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0 | 0 | 0
Not completed — Requirement for Alternative Therapy | 0 | 1 | 0 | 0 | 0
Period: Adjuvant Phase
Arm/Group | ABP 980 | Trastuzumab | ABP 980/ABP 980 | Trastuzumab/Trastuzumab | Trastuzumab/ABP 980
Started | 0 | 0 | 349 (Nine participants discontinued the study after surgery but before entering adjuvant phase.) | 171 (Two participants discontinued the study after surgery but before entering adjuvant phase.) | 171 (Three participants discontinued the study after surgery but before entering adjuvant phase.)
Completed | 0 | 0 | 323 | 164 | 157
Not Completed | 0 | 0 | 26 | 7 | 14
Not completed — Other | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 3
Not completed — Disease Progression or Recurrence | 0 | 0 | 12 | 4 | 3
Not completed — Physician Decision | 0 | 0 | 9 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABP 980 | Trastuzumab | Total
Number analyzed (Participants) | 364 | 361 | 725
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (10.72) | 52.7 (11.29) | 52.7 (11.00)
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 140 | 134 | 274
  ≥ 50 years | 224 | 227 | 451
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 364 | 361 | 725
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 331 | 333 | 664
  Black or African American | 10 | 4 | 14
  Asian | 2 | 3 | 5
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Other | 20 | 21 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 36 | 68
  Not Hispanic or Latino | 332 | 324 | 656
  Not allowed to collect | 0 | 1 | 1
Tumor Stage [Count of Participants; unit: Participants] — In the Tumor Node Metastasis (TNM) staging system, a "T" followed by a number shows the size of the tumor. Less than T4 indicates a tumor that is 5 cm or less. T4 indicates the tumor is any size, but has spread beyond the breast tissue to the chest wall and/or skin.
  Participants
    < T4 | 282 | 281 | 563
    T4 | 82 | 80 | 162
Axilla Lymph Node Involvement [Count of Participants; unit: Participants]
  Yes | 277 | 266 | 543
  No | 87 | 95 | 182
Hormone Receptor Status [Count of Participants; unit: Participants]
  Estrogen and/or progesterone receptor positive | 265 | 268 | 533
  Estrogen and progesterone receptor negative | 99 | 93 | 192
Paclitaxel Dosing Schedule [Count of Participants; unit: Participants]
  Every 3 weeks | 256 | 258 | 514
  Every week | 108 | 103 | 211
Geographic Region [Count of Participants; unit: Participants]
  Eastern Europe | 271 | 273 | 544
  Western Europe | 43 | 46 | 89
  Other | 50 | 42 | 92

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Pathologic Complete Response
Description: Pathologic complete response (pCR) was defined as the absence of invasive tumor cells in the breast tissue and in axillary lymph nodes, regardless of residual ductal carcinoma in situ (DCIS).
  Participants underwent a lumpectomy or mastectomy with sentinel lymph node dissection (SLND) or axillary lymph node dissection (ALND) within 3 to 7 weeks after the last dose of study drug in the neoadjuvant phase. The pathology evaluation of surgical specimens for pCR analysis was conducted by local laboratories at the study sites.
Time Frame: 3 to 7 weeks after the last dose of study drug in the neoadjuvant phase
Population: The pCR evaluable population, which included all randomized participants who received any amount of study drug, underwent the surgery, and had a non-missing evaluable pCR assessment from the local laboratory evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | ABP 980 | Trastuzumab
Number analyzed (Participants) | 358 | 338
percentage of participants | 48.0 | 40.5
Statistical Analysis 1: Comparison: ABP 980 vs Trastuzumab; The clinical equivalence between ABP 980 and trastuzumab was first evaluated by comparing the 2-sided 90% confidence interval (CI) of the Risk Difference (RD; ABP 980 - Trastuzumab) of pCR between ABP 980 and trastuzumab with a fixed margin of (-13%, 13%), estimated using a generalized linear model adjusted for stratification factors tumor (T)-stage, nodal status, hormone receptor status, planned paclitaxel dosing schedule, and geographic region; Test type: Equivalence — The clinical equivalence between ABP 980 and trastuzumab was first evaluated by comparing the 2-sided 90% CI of the risk difference of pCR between ABP 980 and trastuzumab with a fixed margin of (-13%, 13%); p = 0.0508, Generalized linear model; Generalized linear model adjusted for the randomization stratification factors; Risk Difference (RD) = 7.3, 90% CI 2-sided [1.2 to 13.4]
Statistical Analysis 2: Comparison: ABP 980 vs Trastuzumab; If the test of equivalence on the RD of pCR was successful, then equivalence was tested on the Risk Ratio (RR; ABP 980 / Trastuzumab) of pCR at a 2-sided significance level of 0.05 by comparing the 2-sided 90% CI of the RR of pCR between ABP 980 and trastuzumab, estimated using a generalized linear model adjusted for stratification factors: tumor (T)-stage, nodal status, hormone receptor status, planned paclitaxel dosing schedule, and geographic region; Test type: Equivalence — If the test of equivalence on the RD of pCR was successful, then equivalence was tested on the risk ratio of pCR at a 2-sided significance level of 0.05 by comparing the 2-sided 90% CI of the RR of pCR between ABP 980 and trastuzumab estimated using a generalized linear model adjusted for stratification factors, with the margin of (0.7586, 1/0.7586). If the test of equivalence on the RD was not successful, the RR of pCR and 90% CI were considered to be descriptive; p = 0.0430, Generalized linear model; Generalized linear model adjusted for the randomization stratification factors; Risk Ratio (RR) = 1.1877, 90% CI 2-sided [1.0327 to 1.3660]

2. Secondary Outcome: Percentage of Participants With a Pathologic Complete Response in Breast Tissue Only
Description: Pathologic complete response (pCR) was defined as the absence of invasive tumor cells in the breast tissue, regardless of residual ductal carcinoma in situ (DCIS).
  Participants underwent a lumpectomy or mastectomy with sentinel lymph node dissection (SLND) or axillary lymph node dissection (ALND) within 3 to 7 weeks after the last dose of study drug in the neoadjuvant phase. The pathology evaluation of surgical specimens for pCR analysis was conducted by local laboratories at the study sites.
Time Frame: 3 to 7 weeks after the last dose of study drug in the neoadjuvant phase
Population: pCR evaluable population
Measure: Number; unit: percentage of participants
Arm/Group | ABP 980 | Trastuzumab
Number analyzed (Participants) | 358 | 338
percentage of participants | 51.1 | 45.0
Statistical Analysis 1: Comparison: ABP 980 vs Trastuzumab; The analysis of risk difference (ABP 980 - Trastuzumab) estimated using a generalized linear model adjusted for the randomization stratification factors T-stage, node status, hormone receptor status, planned paclitaxel dosing schedule, and geographic region; Test type: Other — Analyses of secondary endpoints were prespecified to be considered descriptive only; p = 0.1086, Generalized linear model; Generalized linear model adjusted for the randomization stratification factors; Risk Difference (RD) = 6.0, 90% CI 2-sided [-0.2 to 12.2]
Statistical Analysis 2: Comparison: ABP 980 vs Trastuzumab; The analysis of risk ratio (ABP 980 / Trastuzumab) estimated using a generalized linear model adjusted for the randomization stratification factors T-stage, node status, hormone receptor status, planned paclitaxel dosing schedule, and geographic region; Test type: Other — Analyses of secondary endpoints were prespecified to be considered descriptive only; p = 0.0807, Generalized linear model; Generalized linear model adjusted for the randomization stratification factors; Risk Ratio (RR) = 1.1463, 90% CI 2-sided [1.0080 to 1.3035]

3. Secondary Outcome: Percentage of Participants With a Pathologic Complete Response in Breast Tissue and Axillary Lymph Nodes and Absence of DCIS
Description: Pathological complete response was defined as the absence of invasive tumor cells in the breast tissue and axillary lymph node(s) and absence of residual DCIS.
  Participants underwent a lumpectomy or mastectomy with sentinel lymph node dissection (SLND) or axillary lymph node dissection (ALND) within 3 to 7 weeks after the last dose of study drug in the neoadjuvant phase. The pathology evaluation of surgical specimens for pCR analysis was conducted by local laboratories at the study sites.
Time Frame: 3 to 7 weeks after the last dose of study drug in the neoadjuvant phase
Population: pCR evaluable population
Measure: Number; unit: percentage of participants
Arm/Group | ABP 980 | Trastuzumab
Number analyzed (Participants) | 358 | 338
percentage of participants | 37.7 | 29.6
Statistical Analysis 1: Comparison: ABP 980 vs Trastuzumab; [analysis description as in outcome 2, analysis 1]; Test type: Other — Analyses of secondary endpoints were prespecified to be considered descriptive only; p = 0.0253, Generalized linear model; Generalized linear model adjusted for the randomization stratification factors; Risk Difference (RD) = 8.0, 90% CI 2-sided [2.1 to 13.9]
Statistical Analysis 2: Comparison: ABP 980 vs Trastuzumab; [analysis description as in outcome 2, analysis 2]; Test type: Other — Analyses of secondary endpoints were prespecified to be considered descriptive only; p = 0.0245, Generalized linear model; Generalized linear model adjusted for the randomization stratification factors; Risk Ratio (RR) = 1.2746, 90% CI 2-sided [1.0673 to 1.5222]

ADVERSE EVENTS:
Time Frame: Neoadjuvant phase: From the first dose of study drug until 30 days after last dose in the neoadjuvant phase or until the start of the adjuvant phase, up to 16 weeks. Adjuvant phase: From the first dose of study drug after surgery until 30 days after last dose; approximately 40 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Neoadjuvant Phase: ABP 980: Participants received ABP 980 at an initial dose of 8 mg/kg over a 90-minute intravenous (IV) infusion, then 6 mg/kg IV infusion every 3 weeks (Q3W) for 3 additional cycles plus 175 mg/m² paclitaxel Q3W for 4 cycles.
- Neoadjuvant Phase: Trastuzumab: Participants received trastuzumab at an initial dose of 8 mg/kg over a 90-minute IV infusion, then 6 mg/kg IV infusion Q3W for 3 additional cycles plus 175 mg/m² paclitaxel Q3W for 4 cycles.
- Adjuvant Phase: ABP 980/ABP 980: After surgery, participants initially randomized to ABP 980 continued to receive ABP 980 at a dose of 6 mg/kg IV infusion Q3W for up to 1 year from the first day of study drug administration in the neoadjuvant phase.
- Adjuvant Phase: Trastuzumab/Trastuzumab: After surgery, participants originally randomized to trastuzumab were re-randomized and continued to receive trastuzumab at a dose of 6 mg/kg IV infusion Q3W for up to 1 year from the first day of study drug administration in the neoadjuvant phase.
- Adjuvant Phase: Trastuzumab/ABP 980: After surgery, participants originally randomized to trastuzumab were re-randomized and switched to receive ABP 980 at a dose of 6 mg/kg IV infusion Q3W for up to 1 year from the first day of study drug administration in the neoadjuvant phase.
Arm/Group | Neoadjuvant Phase: ABP 980 | Neoadjuvant Phase: Trastuzumab | Adjuvant Phase: ABP 980/ABP 980 | Adjuvant Phase: Trastuzumab/Trastuzumab | Adjuvant Phase: Trastuzumab/ABP 980
Serious Adverse Events (participants affected / at risk) | 18/364 | 5/361 | 18/349 | 6/171 | 6/171
Other Adverse Events (participants affected / at risk) | 227/364 | 220/361 | 124/349 | 49/171 | 60/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Phase: ABP 980 (N=364) | Neoadjuvant Phase: Trastuzumab (N=361) | Adjuvant Phase: ABP 980/ABP 980 (N=349) | Adjuvant Phase: Trastuzumab/Trastuzumab (N=171) | Adjuvant Phase: Trastuzumab/ABP 980 (N=171)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Incision site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Drug dispensing error (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound decomposition (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Phase: ABP 980 (N=364) | Neoadjuvant Phase: Trastuzumab (N=361) | Adjuvant Phase: ABP 980/ABP 980 (N=349) | Adjuvant Phase: Trastuzumab/Trastuzumab (N=171) | Adjuvant Phase: Trastuzumab/ABP 980 (N=171)
Anaemia (Blood and lymphatic system disorders) | 40 | 38 | 17 | 7 | 10
Leukopenia (Blood and lymphatic system disorders) | 21 | 16 | 15 | 5 | 8
Neutropenia (Blood and lymphatic system disorders) | 53 | 45 | 25 | 10 | 6
Diarrhoea (Gastrointestinal disorders) | 23 | 19 | 9 | 2 | 4
Nausea (Gastrointestinal disorders) | 21 | 18 | 11 | 3 | 2
Asthenia (General disorders) | 54 | 59 | 17 | 7 | 10
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 37 | 17 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 63 | 55 | 20 | 9 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 29 | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 31 | 2 | 3 | 2
Neuropathy peripheral (Nervous system disorders) | 51 | 43 | 8 | 3 | 2
Paraesthesia (Nervous system disorders) | 17 | 21 | 6 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 25 | 22 | 3 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 23 | 3 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.